CLINICAL TRIAL: NCT00657943
Title: The Effect of Metformin Versus Placebo, Including Three Insulin-Analogue Regimens With Variating Postprandial Glucose Regulation, on CIMT in T2DM Patients - A Randomized, Multicenter Trial
Brief Title: The Copenhagen Insulin and Metformin Therapy Trial
Acronym: CIMT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: Hvidovre University Hospital (Other); Hillerod Hospital, Denmark (Other); Frederiksberg University Hospital (Other); University Hospital, Gentofte, Copenhagen (Other); Rigshospitalet, Denmark (Other); Bispebjerg Hospital (Other); Herlev Hospital (Other); Zealand University Hospital (Other); Copenhagen Trial Unit, Center for Clinical Intervention Research (Other); Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Lise Tarnow, professor, Steno Diabetes Center Copenhagen
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: EudraCT 2007-006665-33
Record Dates: First submitted 2008-04-08; First posted 2008-04-14 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-02

CONDITIONS: Type 2 Diabetes; Atherosclerosis; Arteriosclerosis
Keywords: carotid; intima; media; thickness; insulin; metformin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Atherosclerosis; Arteriosclerosis; Insulin Resistance | interventions — Metformin; Insulin Detemir; Insulin Aspart

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- 1M (Experimental): Metformin + Levemir x1
  Interventions: Drug: metformin; Drug: insulin detemir
- 1P (Placebo Comparator): Placebo + Levemir x1
  Interventions: Drug: insulin detemir
- 2M (Experimental): metformin + NovoMix
  Interventions: Drug: metformin; Drug: insulin aspart + insulin aspart protamin
- 2P (Placebo Comparator): Placebo + NovoMix
  Interventions: Drug: insulin aspart + insulin aspart protamin
- 3M (Experimental): Metformin + 4x therapy
  Interventions: Drug: metformin; Drug: insulin detemir; Drug: Insulin aspart
- 3P (Placebo Comparator): Placebo + 4x therapy
  Interventions: Drug: insulin detemir; Drug: Insulin aspart

INTERVENTIONS:
Drug: metformin — metformin tablets 2 g x 2
  Other Names: glucophage
  Arms: 1M; 2M; 3M
Drug: insulin detemir — insulin as requested
  Other Names: Levemir
  Arms: 1M; 1P; 3M; 3P
Drug: insulin aspart + insulin aspart protamin — insulin as requested
  Other Names: novomix
  Arms: 2M; 2P
Drug: Insulin aspart — insulin as requested
  Other Names: NovoRapid
  Arms: 3M; 3P

SUMMARY:
Type 2 Diabetes Mellitus patients (T2DM) have an increased mortality rate due to macrovascular disease. The primary objective of the study is to evaluate the effect of an 18-month treatment with metformin versus placebo in combination with one of three insulin analogue regimens following a treat-to-target principle. The primary outcome measure is change in wall thickness of the carotic arteries(CIMT)measured by ultrasound. A total of 900 patients with T2DM and HbA1c above 7.5% will be included.

ELIGIBILITY:
Inclusion Criteria:

* Males and females over 30 years of age
* Type 2 diabetes
* Body mass index (BMI): 25.0-39.9 kg/m2
* HbA1c above 7.5 %
* Antidiabetic tablet-treatment during 1 year minimum AND / OR
* Insulin treatment during a minimum of 3 months
* Negative pregnancy test
* Signed, informed consent

Exclusion Criteria:

* MI, coronary revascularization, TCI,or apoplexy within the last 3 months
* TCI with verified stenosis of above 70%
* Heart failure (NYHA class III or IV)
* Former cancer patient, unless disease-free period of more than 5 years
* estimated creatinine clearance < 60 ml/min Liver disease
* Alcohol abuse
* Drug abuse
* Retinopathy with on-going laser treatment at start of study
* Other acute or chronic serious disease leading to hypoxia
* Pregnant or breastfeeding women
* Women of child-bearing potential, not using contraceptives
* Allergy to medication used in the study
* Incapable of understanding the nature of the informed consent

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 415 (Actual)
Dates: Start 2008-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Carotid intima media thickness | 18 months

SECONDARY OUTCOMES:
adverse events | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Almdal, MD DMSc, Principal Investigator — Hvidovre University Hospital
Locations (9):
- Denmark (9):
  - Rigshospitalet, Copenhagen
  - Bispebjerg Hospital, Copenhagen
  - Frederiksberg Hospital, Frederiksberg
  - Gentofte Sygehus, Gentofte Municipality
  - Steno Diabetes Center, Gentofte Municipality
  - Herlev Hospital, Herlev
  - Hillerod Sygehus, Hillerød
  - Hvidovre Hospital, Hvidovre
  - Køge Sygehus, Køge

REFERENCES:
- [Derived] Olsen MH, Almdal TP, Madsbad S, Ovesen C, Gluud C, Sneppen SB, Breum L, Hedetoft C, Krarup T, Lundby-Christensen L, Mathiesen ER, Roder ME, Vestergaard H, Wiinberg N, Jakobsen JC. Quality of life, patient satisfaction, and cardiovascular outcomes of the randomised 2 x 3 factorial Copenhagen insulin and Metformin therapy (CIMT) trial - A detailed statistical analysis plan. Contemp Clin Trials Commun. 2023 Feb 24;33:101095. doi: 10.1016/j.conctc.2023.101095. eCollection 2023 Jun. PMID 36923108
- [Derived] Hansen CS, Lundby-Christiansen L, Tarnow L, Gluud C, Hedetoft C, Thorsteinsson B, Hemmingsen B, Wiinberg N, Sneppen SB, Lund SS, Krarup T, Madsbad S, Almdal T, Carstensen B, Jorgensen ME; CIMT study group. Metformin may adversely affect orthostatic blood pressure recovery in patients with type 2 diabetes: substudy from the placebo-controlled Copenhagen Insulin and Metformin Therapy (CIMT) trial. Cardiovasc Diabetol. 2020 Sep 26;19(1):150. doi: 10.1186/s12933-020-01131-3. PMID 32979921
- [Derived] Nordklint AK, Almdal TP, Vestergaard P, Lundby-Christensen L, Boesgaard TW, Breum L, Gade-Rasmussen B, Sneppen SB, Gluud C, Hemmingsen B, Jensen T, Krarup T, Madsbad S, Mathiesen ER, Perrild H, Tarnow L, Thorsteinsson B, Vestergaard H, Lund SS, Eiken P. The effect of metformin versus placebo in combination with insulin analogues on bone mineral density and trabecular bone score in patients with type 2 diabetes mellitus: a randomized placebo-controlled trial. Osteoporos Int. 2018 Nov;29(11):2517-2526. doi: 10.1007/s00198-018-4637-z. Epub 2018 Jul 19. PMID 30027438
- [Derived] Lundby-Christensen L, Vaag A, Tarnow L, Almdal TP, Lund SS, Wetterslev J, Gluud C, Boesgaard TW, Wiinberg N, Perrild H, Krarup T, Snorgaard O, Gade-Rasmussen B, Thorsteinsson B, Roder M, Mathiesen ER, Jensen T, Vestergaard H, Hedetoft C, Breum L, Duun E, Sneppen SB, Pedersen O, Hemmingsen B, Carstensen B, Madsbad S. Effects of biphasic, basal-bolus or basal insulin analogue treatments on carotid intima-media thickness in patients with type 2 diabetes mellitus: the randomised Copenhagen Insulin and Metformin Therapy (CIMT) trial. BMJ Open. 2016 Feb 25;6(2):e008377. doi: 10.1136/bmjopen-2015-008377. PMID 26916685
- [Derived] Lundby-Christensen L, Tarnow L, Boesgaard TW, Lund SS, Wiinberg N, Perrild H, Krarup T, Snorgaard O, Gade-Rasmussen B, Thorsteinsson B, Roder M, Mathiesen ER, Jensen T, Vestergaard H, Hedetoft C, Breum L, Duun E, Sneppen SB, Pedersen O, Hemmingsen B, Carstensen B, Madsbad S, Gluud C, Wetterslev J, Vaag A, Almdal TP. Metformin versus placebo in combination with insulin analogues in patients with type 2 diabetes mellitus-the randomised, blinded Copenhagen Insulin and Metformin Therapy (CIMT) trial. BMJ Open. 2016 Feb 25;6(2):e008376. doi: 10.1136/bmjopen-2015-008376. PMID 26916684